CLINICAL TRIAL: NCT05366088
Title: Mindfulness-Based Cognitive Therapy (MBCT) vs. Health Enhancement Program (HEP) Active Control for Late-Life Depression: An RCT
Brief Title: RCT of MBCT vs HEP for Late-Life Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Double record
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Principal Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 427282
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Depression in Old Age; Quality of Life
Keywords: Late-life depression; Quality of Life; Mindfulness-Based Cognitive Therapy; Behavioural Activation; Executive Functioning; Processing Speed
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): Online group sessions 90minutes/week, for 8 weeks, and amount of home practice (~30 mins/day, 6 days/week), based on the manualized protocol developed by co-I Dr. Segal and will be delivered by social workers (or equivalent) with ≥3 years of experience delivering MBCT and training for official certification from the Center for Mindfulness Studies (Toronto).
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Health Enhancement Program (Active Comparator): Online group sessions 90minutes/week for 8 weeks, and amount of home practice (~30 mins/day, 6 days/week). HEP will be delivered by social workers (or equivalent) who have received the official training course from HEP's developers at the University of Wisconsin.
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — MBCT is an 8-week therapy integrating formal mindfulness meditation (e.g. breath and body awareness) and informal mindfulness (e.g. eating, walking). Participants are taught to attend non-judgmentally to present moment experiences. MBCT includes cognitive therapy techniques to target the ruminative thought processes and identification with negative emotions seen in depression. MBCT teaches participants how to disengage from habitual ("automatic") dysfunctional cognitive routines, in particular depression-related ruminative thought patterns that perpetuate depressive symptoms and increase vulnerability to relapse.
  Arms: Mindfulness-Based Cognitive Therapy
Behavioral: Health Enhancement Program — HEP teaches health-enhancing techniques and was designed by University of Wisconsin and NIH as a manualized active control group program for mindfulness-based intervention trials (53,54). We have tailored HEP to be structurally equivalent to MBCT. HEP will be delivered by social workers (or equivalent) who have received the official training course from HEP's developers at the University of Wisconsin. Participants will learn about health promotion, healthy diet, music, and gentle exercise, but not about breathing techniques or meditation.
  Arms: Health Enhancement Program

SUMMARY:
Study Design & Recruitment: Phase III randomized controlled trial (RCT) with 100-110 patients. Participants >60 years old, with symptoms of late-life depression (LLD; MADRS score>=10), excluding dementia and other psychiatric comorbidities, will be recruited in Montreal and via social media, across Canada.

Interventions: Mindfulness-based Cognitive Therapy (MBCT) or Health Enhancement Program (HEP) for 8-weeks, in addition to treat as usual (TAU). MBCT and HEP will have the same group sizes, meeting frequency, and amount of home practice. HEP is a recognized active control where participants learn about diet and exercise, but not meditation.

DETAILED DESCRIPTION:
Late life depression (LLD) affects 5 million American seniors yearly with $1.81 billion in direct health-care costs. Biomarkers of LLD have consistently been linked to elevated dementia risk. Mindfulness-based cognitive therapy (MBCT) holds promise for treating symptoms of depression, ameliorating cognitive deficits and preventing decline in older adults by targeting brain circuits implicated in memory and attention. While preliminary findings are promising, the effects of mindfulness delivered through virtual videoconferencing platforms have not been assessed in older adults with depression. This proposed research aims are:

Primary Objective: Using an 8-week RCT, assess whether MBCT improves scores of LLD and quality of life compared to an active control (Health Enhancement Program (HEP)). Hypothesis 1(A): The MBCT group will have a lower score in the Montgomery Asberg Depression Scale (MADRS) at 8-weeks, compared to HEP controls. Hypothesis 1(B): The MBCT group will have higher scores of quality of life (EQ-5D) scores at 8-weeks.

Secondary Objective: To investigate the effects of MBCT on cognitive function in LLD. Hypothesis 2: MBCT will lead to higher scores in executive functioning and processing speed at 8 weeks.

Exploratory Objective: To investigate effects of MBCT on scores of anxiety (GAD-7) and mindfulness presence (Five-Factor Mindfulness Questionnaire (FFMQ) Hypothesis 3(A): The MBCT group will have reduced scores in the Generalized Anxiety Disorder 7 (GAD-7) at 8-weeks, compared to HEP controls. Hypothesis 3(B): The MBCT group will have a higher score in mindfulness presence (FFMQ), compared to HEP controls.

One-hundred (n =100) patients with LLD will be recruited at various centres in Montreal and throughout Canada via social media. Participants will undergo stratified randomization to either MBCT or Health Enhancement Program (HEP) intervention groups. The investigators will assess changes in (1) depression symptoms and quality of life, (2) processing speed and executive functioning, (3) anxiety and mindfulness presence, at baseline (0 weeks), post intervention (8 weeks), after baseline. Raters and clinicians will be blinded to group allocation while participants will be blinded to the study hypotheses.

The proposed study will assess the clinical potential of MBCT to improve symptoms of depression, as well as examine its impact on quality of life and cognition. If virtual delivery of MBCT is found to be effective in treating LLD and improving quality of life, the potential exists to implement this intervention at the study sites, across Canada, and internationally.

ELIGIBILITY:
Inclusion Criteria:

1. MADRS score ≥ 10 (experiencing symptoms of moderate/severe depression) at baseline
2. Ability to provide informed consent (shown as to be able to explain back to the research assistant the purpose of the study as well as voluntary participation, rights, time commitments, etc.)
3. participants who have access to internet and basic digital skills to use their computer/tablet
4. willing and able to attend ≥75% of MBCT or HEP sessions
5. adequate understanding of English or French
6. ability to sit for 90 minutes without discomfort
7. willing to inform if any change is made to their psychotropic medications and dosage for the first 8 weeks of the study

Exclusion Criteria:

1. cognitive deficits at baseline, as defined by MoCA score <19
2. diagnosis of post-traumatic stress disorder, bipolar I or II disorder, primary psychotic disorder (e.g. schizophrenia, schizoaffective disorder), and/or severe personality disorder interfering with ability to function in a group setting intervention on a regular basis
3. substance abuse within the past 6 months
4. high suicide risk (e.g., active suicidal ideation and/or recent intent or plan)
5. significant visual or hearing impairment
6. significant impairments in fine motor skills
7. any medical illnesses that could prevent the participant from engaging in the intervention
8. history of psychiatric hospitalization in the last 3 months

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) score | 8 weeks
  Depression Symptoms, score results suggest mild, moderate or sever depression

SECONDARY OUTCOMES:
Quality of Life 5 dimensions | 8 weeks
  is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored on a 5-level severity ranking that ranges from "no problems" through "extreme problems."

OTHER OUTCOMES:
executive functioning and processing speed | 8 weeks
  outcome measures on cognition (Processing speed: Trails Making Test A and WAIS-IV Digit Symbol, and executive functioning: Trails Making Test B, WAIS- IV Digit Span, and Verbal Fluency Test)
anxiety, Mindfulness Presence and global cognition | 8 weeks
  Exploratory outcomes measured by the following scales: anxiety (Generalized Anxiety Disorder 7: GAD-7), Mindfulness Presence (FFMQ) and global cognition (Montreal cognitive assessment, MoCA)

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Davis Institute, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bein M, Lesage M, Dikaios E, Chakravarty M, Segal Z, Royal I, Speechley M, Schiavetto A, Blumberger D, Sacchet MD, Therriault J, Gruber J, Tourjman V, Richard-Devantoy S, Nair V, Bruneau MA, Rej S, Lifshitz M, Sekhon H. Mindfulness-based cognitive therapy vs. a health enhancement program for the treatment of late-life depression: Study protocol for a multi-site randomized controlled trial. Front Aging Neurosci. 2022 Sep 1;14:976636. doi: 10.3389/fnagi.2022.976636. eCollection 2022. PMID 36118690